CLINICAL TRIAL: NCT01149837
Title: In Vitro Diagnostic Study for Supplemental Testing of Anti-HTLV-I/II Reactive Human Blood Specimens
Brief Title: Evaluation of InnoLIA HTLV I/II Score
Status: Completed | Type: Observational
Sponsor: Creative Testing Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: BB-IND 14309
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Human T-Lymphotrophic Virus Type I and/or Type II
Keywords: HTLV; HTLV I; HTLV II; HTLV Type I and/or HTLV Type II antibody

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human serum and/or human plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- residual blood donor samples: Protocol describes testing an HTLV-I/II antibody reactive population from this cohort using the InnoLIA HTLV I/II Score line immunoassay
  Interventions: Device: InnoLIA HTLV I/II Score line immunoassay

INTERVENTIONS:
Device: InnoLIA HTLV I/II Score line immunoassay — This intervention consists of testing a residual serum or plasma sample from a blood donation or donor follow-up sample using the InnoLIA HTLV I/II Score line immunoassay

SUMMARY:
The InnoLIA HTLV I/II Score is an in vitro diagnostic test for confirmation of antibodies to human T-cell lymphotropic virus (HTLV) type I and type II in human blood samples. It is intended as a supplemental test for blood donor samples that are reactive in routine anti-HTLV screening tests. This study will determine if the test is useful for donor counseling purposes.

DETAILED DESCRIPTION:
The InnoLIA HTLV I/II Score study consists of three sub-studies. The first sub-study will determine the sensitivity, specificity and accuracy of HTLV type assignment using well-characterized samples from the NIH-funded HTLV Outcomes Study (HOST). The second sub-study will compare automated reading and interpretation of test results with manual reading and interpretation using a sub-set of samples tested in the initial study. The third sub-study allows for use of the InnoLIA HTLV I/II Score as a supplemental test for whole blood and HCT/P donors testing repeatedly reactive with an FDA-approved donor screening test for anti-HTLV-I/II.

ELIGIBILITY:
Inclusion Criteria:

* Subjects completing a health history evaluation for routine donor screening
* Subjects willing and able to provide informed consent
* Subjects testing repeat reactive on a licensed screening test for HTLV antibodies

Exclusion Criteria:

* Subjects not meeting health history criteria for routine donor screening
* Subjects unwilling and unable to provide informed consent
* Subjects testing negative on a licensed screening test for HTLV antibodies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Whole blood and HCT/P donor samples found repeatedly reactive for anti-HTLV-I/II using an FDA approved donor screening test
Sampling Method: Probability Sample
Enrollment: 3305 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
INNO-LIA HTLV I/II Score Testing | September 2013 through December 2013, up to 3 months
  322 residual donor samples tested
INNO-LIA HTLV I/II Score Testing | January 2014 through December 2014, up to one year
  896 residual donor samples tested
INNO-LIA HTLV I/II Score Testing | January 2015 through December 2015, up to one year
  630 residual donor samples tested
INNO-LIA HTLV I/II Score Testing | January 2016 through May 2016
  315 residual donor samples tested

CONTACTS AND LOCATIONS:
Overall Officials: Phillip C Williamson, PhD, Principal Investigator — Creative Testing Solutions
Locations (1):
- Creative Testing Solutions, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided